CLINICAL TRIAL: NCT02716532
Title: Bioavailability of Medium Chain Triglycerides (MCTs) in Comatose Patients With Acute Brain Injury (ABI)
Acronym: MCTs and ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15.03.CLI
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Injuries, Acute Brain; Severe Trauma Brain Injury (sTBI); Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptamen AF (Other): over 7 days
  Interventions: Dietary Supplement: Peptamen AF

INTERVENTIONS:
Dietary Supplement: Peptamen AF — Each patient will receive Peptamen AF throughout the trial.

SUMMARY:
This study will be targeting patients suffering from acute brain injury (ABI), including those with severe trauma brain injury (sTBI) and those with aneurysmal sub arachnoid hemorrhage (aSAH).

This clinical study is an open-label, non-randomized, single-center, exploratory metabolic study.

The primary objective is to determine changes from baseline (before enteral administration of Peptamen AF) in plasma and brain extracellular levels of MCFAs and Ketone bodies in sTBI patients upon Peptamen AF nutritional support.

ELIGIBILITY:
Inclusion Criteria:

* Comatose patients (defined by an initial Glasgow Coma Scale (GCS) < 9) following sTBI or aSAH.
* Female or male, aged >18.
* Abnormal head CT-Scan (contusions, hematoma).
* Intracranial monitoring with CMD, [PbtO2] and [ICP] probes as part of standard of care.
* Written informed consent from an independent physician (not associated to the research project) who provides medical follow-up and defends patient's interests.
* Written informed consent from patient relative/legal representative confirming the presumed patient willingness to participate in the study

Exclusion Criteria:

* Signs of brain death or expected brain death within 48h.
* Pregnancy.
* Hemodynamic instability (circulatory shock, requiring vasopressors).
* Renal or liver insufficiency .
* Chronic intestinal disease.
* Patients requiring parenteral nutrition .
* Currently participating or having participated in another clinical trial during the month preceding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline of plasma and brain extracellular (CMD fluid) levels of MCFAs and KBs in sTBI upon Peptamen AF nutritional support | Over 7 days

SECONDARY OUTCOMES:
Changes from baseline of plasma and brain extracellular levels of MCFAs and KBs in aSAH patients | After at least 2 consecutive days of stable enteral nutrition
Change from baseline in plasma and brain extracellular levels of MCFAs and KBs in all patients | Over 7 days (not necessarily at stable EN).
As part of standard care, monitoring of intra-cerebral physiologic and metabolic variables and correlation with brain MCFAs and KBs levels in all patients | Over 7 days
Changes from baseline in cerebrospinal fluid of MCFAs and KBs concentrations in all patients with extra-ventricular drainage (EVD) as part of standard care | Over 7 days
To correlate MCFAs and KBs levels in CMD, plasma and cerebral spinal fluid in all patients | Over 7 days
Evaluation of the time to reach two days of stable nutrition in all patients | Over 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cuénoud, PhD, Study Director — Nestec SA
Locations (1):
- Department of Intensive Care Medicine CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No